CLINICAL TRIAL: NCT02876224
Title: A Phase Ib Open-Label Study Evaluating the Safety, Tolerability and Pharmacokinetics of Cobimetinib in Combination With Bevacizumab and Immunotherapy When Administered in Patients With Gastrointestinal and Other Tumors
Brief Title: Study of Cobimetinib in Combination With Atezolizumab and Bevacizumab in Participants With Gastrointestinal and Other Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: CO39083; 2016-000584-16 (EudraCT Number)
Record Dates: First submitted 2016-08-18; First posted 2016-08-23 (Estimated); Last update posted 2019-08-13 (Actual); Status verified 2019-08

CONDITIONS: Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms | interventions — atezolizumab; Bevacizumab; cobimetinib

ARMS (3):
- Cobimetinib + Bevacizumab + Atezolizumab (Stage 1: SRP) (Experimental): Stage 1 Safety Run-in Phase (SRP): Approximately 12 participants will receive cobimetinib 60 milligrams (mg) orally once daily for Days 1-21 with atezolizumab 840 mg and bevacizumab 5 milligrams per kilogram (mg/kg) administered by IV infusion on Days 1 and 15 of each 28-day cycle. Atezolizumab will be administered first, followed by bevacizumab, with a minimum of 60 minutes between dosing. Upon determination of the safety and tolerability of the treatment regimen, the study will proceed to Stage 2: dose expansion phase. If the results from the safety run-in phase require dose reduction in cobimetinib, then an additional Stage 1 cohort will be opened. Treatment will continue until the participant has disease progression according to Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST v1.1), unacceptable toxicity, death, participant or physician decision to withdraw, or pregnancy, whichever occurs first.
  Interventions: Drug: Atezolizumab; Drug: Bevacizumab; Drug: Cobimetinib
- Cobimetinib + Bevacizumab + Atezolizumab (Stage 2: BC) (Experimental): Stage 2 Biopsy Cohort (BC): Approximately 7 evaluable participants in the biopsy cohort in expansion phase will receive bevacizumab 5 mg/kg IV on Cycle 1 Days 1 and 15 (tumor biopsy on Cycle 1 Day 8) and cobimetinib (at dose determined during safety run-in phase) orally on Cycle 1 Day 15 to Cycle 2 Day 14 (tumor biopsy on Cycle 1 Day 22). From Cycle 2 onwards, participants will follow the same treatment regimen for bevacizumab and atezolizumab (optional tumor biopsy on Cycle 2 Day 22) as those in the safety run-in phase and expansion cohort, and for cobimetinib cycles start at Day 15 and will continue 21 days to Day 7 of next cycle. Atezolizumab will be administered first, followed by bevacizumab, with a minimum of 60 minutes between dosing. Biopsies must be collected before the initiation of cobimetinib and atezolizumab. Treatment will continue until disease progression according to RECIST v1.1, unacceptable toxicity, death, decision to withdraw, or pregnancy, whichever occurs first.
  Interventions: Drug: Atezolizumab; Drug: Bevacizumab; Drug: Cobimetinib
- Cobimetinib + Bevacizumab + Atezolizumab (Stage 2: EC) (Experimental): Stage 2 Expansion Cohort (EC): Approximately 14 participants will receive cobimetinib (at dose determined during safety run-in phase) orally once daily for Days 1-21 with atezolizumab 840 mg and bevacizumab 5 mg/kg administered by IV infusion on Days 1 and 15 of each 28-day cycle. Atezolizumab will be administered first, followed by bevacizumab, with a minimum of 60 minutes between dosing. Treatment will continue until the participant has disease progression according to RECIST v1.1, unacceptable toxicity, death, participant or physician decision to withdraw, or pregnancy, whichever occurs first.
  Interventions: Drug: Atezolizumab; Drug: Bevacizumab; Drug: Cobimetinib

INTERVENTIONS:
Drug: Atezolizumab — Atezolizumab 840 mg will be administered by IV infusion on Days 1 and 15 of each 28-day cycle.
  Other Names: RO5541267
Drug: Bevacizumab — Bevacizumab 5 mg/kg will be administered by IV infusion on Days 1 and 15 of each 28-day cycle.
  Other Names: RO4876646
Drug: Cobimetinib — Cobimetinib 60 mg or at dose determined during safety run-in phase will be administered orally once daily for 21 days of each 28-day cycle as specified in the arm descriptions.
  Other Names: RO5514041

SUMMARY:
This is an open-label, multicenter, single-arm, two-stage, Phase Ib study designed to assess the safety, tolerability, and pharmacokinetics of oral cobimetinib with intravenous (IV) atezolizumab and bevacizumab in participants with metastatic colorectal cancer (mCRC) who have received and progressed on at least one prior line of therapy that contained a fluoropyrimidine and oxaliplatin or irinotecan. There are two stages in this study: Stage 1 (safety run-in phase) and Stage 2 (dose expansion phase with two cohorts, an expansion cohort and a biopsy cohort).

ELIGIBILITY:
Inclusion Criteria:

* Eastern Cooperative Oncology Group performance status of 0 or 1
* Histologically confirmed unresectable metastatic colorectal adenocarcinoma
* Life expectancy at least 12 weeks
* Progression on a prior line of therapy that contained a fluoropyrimidine and oxaliplatin or irinotecan for unresectable metastatic colorectal adenocarcinoma
* Measurable disease per RECIST v1.1
* Adequate hematologic and end organ function
* Creatinine clearance greater than or equal to (>=) 30 milliliters per minute (mL/min)
* For biopsy cohort, participants must be bevacizumab naive or received the last bevacizumab treatment at least 12 months prior to Cycle 1 Day 1 and according to the investigator's judgment the planned biopsies would not expose participants to substantially increased risk of complications
* For women of childbearing potential, agreement to remain abstinent (refrain from heterosexual intercourse) or use of contraceptive methods that result in a failure rate of less than (<) 1 percent (%) per year during the treatment period and for at least 180 days after the last study treatment
* For men, agreement to remain abstinent (refrain from heterosexual intercourse) or use contraceptive measures, and agreement to refrain from donating sperm

Exclusion Criteria:

* More than one prior line of systemic therapy for advanced CRC
* Participants with known microsatellite (MSI)-high status
* Major surgery or significant traumatic injury within 60 days prior to enrollment
* Minor surgical procedure within 15 days of study Cycle 1 Day 1
* Untreated central nervous system (CNS) metastases
* Treatment with any investigational agent or approved therapy within 28 days
* Malignancies other than colorectal cancer within 5 years prior to Cycle 1 Day 1
* Prior radiation therapy within 30 days prior to study Cycle 1 Day 1 and/or persistence of radiation-related adverse effects
* Prior allogeneic bone marrow transplantation or solid organ transplant for another malignancy in the past
* Spinal cord compression not definitively treated with surgery and/or radiation
* Uncontrolled pleural effusion, pericardial effusion, or ascites requiring recurrent drainage procedures
* Current or recent use of therapeutic oral or parenteral anticoagulants or thrombolytic agents
* Intake of St. John's wort or hyperforin (potent cytochrome P450 [CYP] 3A4 enzyme inducer) or grapefruit juice (potent CYP3A4 enzyme inhibitor) within 7 days prior to initiation of study treatment
* History of severe allergic, anaphylactic, or other hypersensitivity reactions to chimeric or humanized antibodies or fusion proteins
* Known hypersensitivity or allergy to biopharmaceuticals produced in Chinese hamster ovary cells or any components of cobimetinib, atezolizumab, or bevacizumab formulations
* Prior treatment with clusters of differentiation (CD) 137 (CD137) agonists or immune checkpoint blockage therapies, anti-programmed death protein-1, anti-program death-ligand 1, mitogen-activated protein kinase (MEK) inhibitor
* Proteinuria value > 1.0 g at screening
* Uncontrolled glaucoma with intraocular pressure ≥ 21 mmHg
* Hyperglycemia (fasting) ≥ Grade 2
* Human Immunodeficiency Virus (HIV) infection
* Active hepatitis B or hepatitis C
* History of autoimmune disease, clinically significant cardiac or pulmonary dysfunction
* Administration of a live, attenuated vaccine within 4 weeks prior to Cycle 1 Day 1 or at any time during the study and for at least 5 months after the last dose of study drug
* History of or evidence of retinal pathology on ophthalmologic examination that is considered a risk factor for neurosensory retinal detachment/central serous chorioretinopathy, retinal vein occlusion, or neovascular macular degeneration
* History of idiopathic pulmonary fibrosis, organizing pneumonia, drug-induced pneumonitis, or idiopathic pneumonitis
* Uncontrolled tumor pain

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2016-09-30 (Actual); Primary Completion 2019-06-25 (Actual); Study Completion 2019-06-25 (Actual)

PRIMARY OUTCOMES:
Percentage of Participants with Adverse Events | Baseline up to approximately 12 months

SECONDARY OUTCOMES:
Plasma Maximum Concentration (Cmax) of Cobimetinib | Safety run-in phase and expansion cohort: Predose (0 hours) on Cycle 1 Day 15 and Cycle 3 Day 15; 2 to 4 hours postdose on Cycle 1 Day 1 and Cycle 3 Day 15. Biopsy cohort: 0-2 hours predose and 2-4 hours postdose on Cycle 2 Day 1. Each cycle is 28 days.
Plasma Minimum Concentration (Cmin) of Cobimetinib | Safety run-in phase and expansion cohort: Predose (0 hours) on Cycle 1 Day 15 and Cycle 3 Day 15; 2 to 4 hours postdose on Cycle 1 Day 1 and Cycle 3 Day 15. Biopsy cohort: 0-2 hours predose and 2-4 hours postdose on Cycle 2 Day 1. Each cycle is 28 days.
Serum Cmax of Atezolizumab | Baseline up to approximately 12 months (detailed sample collection timepoints are provided in outcome measure description field)
  Safety run-in phase and expansion cohort: Prior to the infusion (0 hours) on Day 1 of Cycles 1, 2, 4, 8, every 8 cycles thereafter (maximum up to 12 months) and on Day 15 of Cycle 3; 30 minutes after end of infusion (infusion duration 30-60 minutes) on Cycle 1 Day 1 and Cycle 3 Day 15; at treatment discontinuation visit (up to 12 months). Biopsy cohort: prior to the infusion (0 hours) on Day 1 of Cycles 3, 5, 9, every 8 cycles thereafter (maximum up to 12 months) and on Day 15 of Cycle 4; 30 minutes after end of infusion on Day 15 of Cycle 4; at treatment discontinuation visit (up to 12 months). Each cycle is 28 days.
Serum Cmin of Atezolizumab | Baseline up to approximately 12 months (detailed sample collection timepoints are provided in outcome measure description field)
  Safety run-in phase and expansion cohort: Prior to the infusion (0 hours) on Day 1 of Cycles 1, 2, 4, 8, every 8 cycles thereafter (maximum up to 12 months) and on Day 15 of Cycle 3; 30 minutes after end of infusion (infusion duration 30-60 minutes) on Cycle 1 Day 1 and Cycle 3 Day 15; at treatment discontinuation visit (up to 12 months). Biopsy cohort: prior to the infusion (0 hours) on Day 1 of Cycles 3, 5, 9, every 8 cycles thereafter (maximum up to 12 months) and on Day 15 of Cycle 4; 30 minutes after end of infusion on Day 15 of Cycle 4; at treatment discontinuation visit (up to 12 months). Each cycle is 28 days.
Serum Cmin of Bevacizumab | Safety run-in phase and expansion cohort: prior to the infusion (0 hours) on Cycle 3 Day 15. Biopsy cohort: prior to the infusion (0 hours) on Cycle 3 Day 1. Each cycle is 28 days.
Percentage of Participants with Anti-therapeutic Antibodies (ATAs) Response to Atezolizumab | Baseline up to approximately 12 months (detailed sample collection timepoints are provided in outcome measure description field)
  Safety run-in phase and expansion cohort: Prior to the infusion (0 hours) on Day 1 of Cycle 1, 2, 4, 8, and every 8 cycles thereafter (maximum up to 12 months) and on Day 15 of Cycle 3; 30 minutes after end of infusion (infusion duration 30-60 minutes) on Cycle 3 Day 15; at treatment discontinuation visit (up to 12 months). Biopsy cohort: prior to the infusion (0 hours) on Day 1 of Cycles 3, 5, 9, every 8 cycles thereafter (maximum up to 12 months) and on Day 15 of Cycle 4; 30 minutes after end of infusion on Day 15 of Cycle 4; at treatment discontinuation visit (up to 12 months). Each cycle is 28 days.

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (6):
- United States (4):
  - University Of Colorado, Aurora, Colorado
  - Memorial Sloan-Kettering Cancer Center, New York, New York
  - Sarah Cannon Research Inst., Nashville, Tennessee
  - The University of Texas MD Anderson Cancer Center, Houston, Texas
- Spain (2):
  - Hospital Universitario Vall d'Hebron, Barcelona
  - START Madrid. Centro Integral Oncologico Clara Campal; CIOCC, Madrid